CLINICAL TRIAL: NCT04649346
Title: The Difference of Oropharyngeal Leak Pressure and Sealing Pressure Between New Supraglottic Airway Devices
Acronym: SGA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907019RINC
Record Dates: First submitted 2020-10-07; First posted 2020-12-02 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-10

CONDITIONS: Oropharyngeal Leak Pressure
Keywords: Supraglottic airway (SGA) devices

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SGA type 1: Observe the function of SGA type 1
- SGA type 2: Observe the function of SGA type 2

SUMMARY:
The difference of oropharyngeal leak pressure and sealing pressure between new supraglottic airway devices.

DETAILED DESCRIPTION:
In this clinical study, investigators want to discuss the issue that oropharyngeal leak pressure and sealing condition with different SGA including air-Q、i-gel、LMA-supreme、AMBU auragain 、ProSeal LMA and other new SGAs.

In the perioperative period, investigators documented respiratory function data including oropharyngeal leak pressure and peak airway pressure in these randomly selected SGA. Oropharyngeal leak pressure was measured by closing the expiratory valve of the circle system at fixed O2 flow 3L/min and noting the airway pressure at which the dial on a calibrated aneroid manometer reached equilibrium.

investigators wanted to compared the respiratory function between air-Q、i-gel、LMA-supreme、AMBU auragain、ProSeal LMA and other new SGAs during surgery and postoperative care unit.

ELIGIBILITY:
Inclusion criteria:

1. 20-80 years old.
2. ASA physical status I or II .
3. Without major organ dysfunction like heart, liver, brain, lung, kidney function failure.

Exclusion criteria:

1. BMI> 35 kg/m2.
2. Risk of aspiration(NPO clear water> 2 hours, solid foods > 8 hours).
3. Difficult airway like head and neck tumor or airway tumor.
4. Limited mouth opening (<2cm).
5. major organ dysfunction including heart, liver, brain, lung, kidney function failure.
6. Major surgery including open heart surgery, laparotomy general surgery, open chest surgery.

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All general anesthesia patients who use SGA.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Oropharyngeal leak pressures | 10 minutes
  oropharyngeal leak pressure units ( cmH2O )

SECONDARY OUTCOMES:
1. The participant's head and neck position 2. The number of attempts required for SGA insertion 3. Ease of gastric tube placement 4. The ventilation score | 180 minutes
  1. The participant's head and neck position (neutral/extension/flexion/rotation)
  2. The number of attempts required for SGA insertion (1/2/3/tracheal intubation)
  3. Ease of gastric tube placement (success/failure/Leak)
  4. The ventilation score was scored from 0 to 3 based on three criteria:
  (1) No leakage with an airway pressure of > 15 cm H2O (2) Bilateral chest excursions with a peak inspiratory pressure of > 20 cm H2O (3) A Square Wave Capnography with each item scoring 0 or 1 point. Thus, if all three criteria were satisfied, the ventilation score was 3.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Chih Min, Principal Investigator — visiting staff
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan